CLINICAL TRIAL: NCT02028793
Title: Factors Related to Work Pressure and Turnover Intention for Pharmacists With Home Pharmaceutical Care
Brief Title: Work Pressure for Pharmacist With Home Pharmaceutical Care
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VGHTCPHARM2
Record Dates: First submitted 2013-11-24; First posted 2014-01-07 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Pressure Factors; Work Load.; Intention of Leaving the Service
Keywords: Pharmaceutical Care, Taiwan, pharmacist, Workload, pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacists provide pharmaceutical care: The group is the community pharmacists who attend the protocol to provide home visit to the patients with heavy health expenditure, through pharmaceutical care approach.

SUMMARY:
National Health Insurance Administration, Taiwan has provided a protocol for community pharmacist to offer home pharmaceutical care for the patients with high health expenditures. Since community pharmacists need to visit patients for consultation and check their medications, it has been thought to have pressure for them in various areas. This study intends to investigate the factors related to the pressure and intention for leaving this protocol. The hypothesis are that community pharmacist who works longer, has economic pressure, and longer year of practice will have higher pressure and strong intention for leaving.

ELIGIBILITY:
Inclusion Criteria:

* community pharmacists who attend the protocol.

Exclusion Criteria:

* community pharmacists who attend any other home pharmaceutical care projects (any types).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community pharmacists who attend the protocol (offered by National Health Insurance Administration,, Taiwan). the protocol is designed to provide home pharmaceutical care (PC) to the patients with heavy health expenditure. This group of community pharmacists needs to operate their pharmacy while offering PC with small amount of payment. This study investigates the work load, pressure, and intention of leaving the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
intention to leave the service | up to four months
  community pharmacist who provides the service will have chance to fill the questionnaire. the major outcome will be his/her intention to leave the service.

SECONDARY OUTCOMES:
work pressure | up to four months
  each community pharmacist will be asked through questionnaire regarding their work pressure related to the pharmaceutical care.
work load | up to four months
  each community pharmacist attends the study will provide what they though about the loading in offering pharmaceutical care.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Shyong Liou, PhD, Principal Investigator — Taichung Veteran General Hospital, Taiwan
Locations (1):
- Community Pharmacies, All Cities in Taiwan, Taiwan, Taiwan

REFERENCES:
- [Background] Folkman S. Personal control and stress and coping processes: a theoretical analysis. J Pers Soc Psychol. 1984 Apr;46(4):839-52. doi: 10.1037//0022-3514.46.4.839. PMID 6737195
- [Background] Mott DA, Doucette WR, Gaither CA, Pedersen CA, Schommer JC. Pharmacists' attitudes toward worklife: results from a national survey of pharmacists. J Am Pharm Assoc (2003). 2004 May-Jun;44(3):326-36. doi: 10.1331/154434504323063968. PMID 15191243
- [Background] Mak VS, March GJ, Clark A, Gilbert AL. Why do Australian registered pharmacists leave the profession? a qualitative study. Int J Clin Pharm. 2013 Feb;35(1):129-37. doi: 10.1007/s11096-012-9720-5. Epub 2012 Oct 30. PMID 23109069
- [Background] Strachota E, Normandin P, O'Brien N, Clary M, Krukow B. Reasons registered nurses leave or change employment status. J Nurs Adm. 2003 Feb;33(2):111-7. doi: 10.1097/00005110-200302000-00008. PMID 12584464
- [Background] Williams LJ, & Hazer, J.T.. Antecedents and consequences of satisfaction and commitment in turnover models: A reanalysis using latent variable structural equation methods. . Journal of Applied Psychology. 1986;71:219-231.
- [Background] Mosadeghrad AM, Ferlie E, Rosenberg D. A study of relationship between job stress, quality of working life and turnover intention among hospital employees. Health Serv Manage Res. 2011 Nov;24(4):170-81. doi: 10.1258/hsmr.2011.011009. PMID 22040944
- [Background] Ramalho de Oliveira D, Brummel AR, Miller DB. Medication therapy management: 10 years of experience in a large integrated health care system. J Manag Care Pharm. 2010 Apr;16(3):185-95. doi: 10.18553/jmcp.2010.16.3.185. PMID 20331323
- [Background] Zarowitz BJ, Stebelsky LA, Muma BK, Romain TM, Peterson EL. Reduction of high-risk polypharmacy drug combinations in patients in a managed care setting. Pharmacotherapy. 2005 Nov;25(11):1636-45. doi: 10.1592/phco.2005.25.11.1636. PMID 16232025